CLINICAL TRIAL: NCT02857062
Title: An Open Label, In-use Tolerance Study in Babies and Children With Dry/Atopic and Very Dry/Atopic Skin, to Evaluate the Acceptability and Skin Tolerability of E45 Eczema Repair Emollient for the Treatment of Atopic or Eczema Prone Skin
Brief Title: To Evaluate the in Use Tolerance of E45 Eczema Repair Emollient in Babies and Children With (Very(Dry/Atopic Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Intertek (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09224-02
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-01

CONDITIONS: Atopic Dermatitis / Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: Open label, in use tolerance study in babies and children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E45 Eczema Repair Emollient (Experimental): Open label, single arm study to evaluate the skin tolerance of E45 Eczema Repair Emollient in babies and children
  Interventions: Device: E45 Eczema Repair Emollient

INTERVENTIONS:
Device: E45 Eczema Repair Emollient — E45 Eczema Repair Emollient

SUMMARY:
The investigation will evaluate, under dermatological control, the cutaneous in-use tolerance of E45 Eczema Repair Emollient with two or three times daily application, over a period of two weeks on children and babies with dry/atopic and very dry/atopic skin.

DETAILED DESCRIPTION:
The investigation is an open label, in-use cutaneous tolerance investigation in children and babies with dry/atopic and very dry/atopic skin, to evaluate the acceptability and skin tolerability of E45 Eczema Repair Emollient.

The investigation will be an 'at home' user investigation where the test product will be applied by the parent/legal guardian to a pre-defined test site (arm or leg) between 2 to 3 times daily, consecutively for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. be female or male
2. be a child aged from ≥3 years to < 12 years or a baby aged from ≥3 months to < 36 months at screening
3. be phototype I - IV (Fitzpatrick Phototyping Scale)
4. have skin that is dry/atopic or very dry/atopic (confirmed by the Dermatologist in consultation with the parent/legal guardian)
5. have mild atopic eczema (as confirmed by the Dermatologist in consultation with the parent/legal guardian) but not undergoing steroid treatment for the condition
6. have only few or no pigmentation on the selected test site
7. be in general good health and mental condition

   In addition the parent/legal guardian must:
8. Both parents in case of shared custody/legal guardian will provide written informed consent for their child/baby to participate in the investigation (children aged 6 years and above, capable of understanding the investigation after it has been explained to them, will be asked to provide assent. Pre-schoolers (2-5 years) will be allowed to express a level of assent verbally relating to their ability to do so)
9. agree to attend the investigation centre, with the child/baby, on the predefined days
10. be willing and capable to follow the investigation requirements

Exclusion Criteria:

1. have chronic or acute skin diseases, except atopic eczema on any part of the body
2. have an active flare up of atopic eczema on any sites of the body at screening
3. known allergy or sensitivity to cosmetic products and/or any ingredients of the investigational product.
4. any systemic illness that would impact on the subjects safety or wellbeing and/or affect the response of the skin or the interpretation of the test results at screening (Day -14 to -7)
5. receiving the following topical or systemic treatments at baseline (Day 0);

   * anti-inflammatory and/or anti-histamines during the previous week
   * cough suppressants and/or topical or inhaled corticosteroids during the previous 2 weeks
   * retinoids and/or immunosuppressants during the previous 6 months
6. have diabetes, acute cardiac and circulatory diseases, HIV, hepatitis
7. participation in other studies/investigations on any part of the body during the last 4 weeks
8. use of dermatological therapeutics on the body within 7 days prior to baseline (Day 0) (use of such products on the face, trunk, hands and nappy area is permitted)
9. swimming within 48 hours prior to baseline (Day 0)
10. intensive/prolonged exposure to the sun within 30 days prior to screening
11. planned changes to subject's diet during the investigation (e.g. weaning)
12. subjects whose parent/legal guardian are employees or who work for a manufacturer of personal care products or for the testing facility
13. subjects in protective care
14. subjects whose parent/legal guardian (who will be applying the investigation product) is allergic to the investigation device ingredients
15. Any clinically significant and relevant abnormalities of medical history and/or any condition or medication that would impact on the subject safety or well-being and/or affect the response of the skin or the interpretation of the test results in the opinion of the Principal Investigator or designee

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Cutaneous Tolerance | 14 Days
  The total irritancy score (Erythema score + Oedema score + Papules score + Vesicles score) for each subject from baseline to end of study as observed by the investigation Dermatologist.
Parental Assessment of Cutaneous Tolerance | 14 Days
  The dermatologist will ask the parent/legal guardian to provide their assessment of tolerance by asking the parent/legal guardian if they considered the product to be well tolerated by their child/baby's skin
Global Assessment of Cutaneous Tolerance | 14 Days
  The dermatologist will make a 'global assessment' of tolerance for each subject based on reported product use/compliance

IPD SHARING:
Plan to Share IPD: No